CLINICAL TRIAL: NCT02473042
Title: Intraoperative Electrical Stimulation of the Acupoint P6 to Prevent Post-Operative Nausea and Vomiting in Women Undergoing Breast Cancer Surgery
Brief Title: Intraoperative Acupoint Stimulation to Prevent Post-Operative Nausea and Vomiting (PONV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2015-0170; NCI-2015-01519 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Post-Operative Nausea and Vomiting; Breast Cancer
Keywords: Post-operative nausea and vomiting; PONV; Breast cancer; Neuromuscular blockade monitor; NMBM; Breast cancer surgery; Prophylactic anti-emetics; Electrical stimulation; Zofran; Ondansetron; Dexamethasone; Decadron; Phenergan; Promethazine; Phenazine; Phencen; Prometh; Prorex; V-Gan; Pepcid; Famotidine; Questionnaire; Survey
MeSH Terms: conditions — Vomiting; Breast Neoplasms; Postoperative Nausea and Vomiting | interventions — Electric Stimulation; Ondansetron; Dexamethasone; Calcium Dobesilate; Promethazine; phenazine; Diphenhydramine; Famotidine; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Electrical Stimulation + Standard of Care Antiemetics (Experimental): Participants receive light electrical stimulation to the wrist area during surgery. Participants also receive standard of care drugs to reduce post-operative nausea and vomiting (PONV).
  Questionnaire completed about participant's pre-treatment expectations and their nausea about 15 minutes after they wake up after surgery, then every 30 minutes until they leave the clinic.
  Interventions: Procedure: Electrical Stimulation; Drug: Zofran; Drug: Dexamethasone; Drug: Phenergan; Drug: Pepcid; Behavioral: Questionnaire
- Standard of Care Antiemetics (Active Comparator): Participants receive standard of care drugs to reduce post-operative nausea and vomiting (PONV).
  Questionnaire completed about participant's pre-treatment expectations and their nausea about 15 minutes after they wake up after surgery, then every 30 minutes until they leave the clinic.
  Interventions: Drug: Zofran; Drug: Dexamethasone; Drug: Phenergan; Drug: Pepcid; Behavioral: Questionnaire

INTERVENTIONS:
Procedure: Electrical Stimulation — Electrical stimulation to the wrist initiated at 1mHz, 1 pulse/second using two leads on a nerve stimulator. Stimulation continued throughout the breast surgery.
  Arms: Electrical Stimulation + Standard of Care Antiemetics
Drug: Zofran — 4 mg by vein for 1 dose.
  Other Names: Ondansetron
Drug: Dexamethasone — 10 mg by vein for 1 dose.
  Other Names: Decadron
Drug: Phenergan — 6.25 mg by vein for 1 dose.
  Other Names: Promethazine; Phenazine; Phencen; Prometh; Prorex; V-Gan
Drug: Pepcid — 10 mg by vein for 1 dose.
  Other Names: Famotidine
Behavioral: Questionnaire — Questionnaire completed about 15 minutes after participant wakes up after surgery, then every 30 minutes until they leave the clinic. It should take about 2 - 3 minutes to complete the questionnaire.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to learn if light electrical stimulation to the wrist area during surgery is feasible in women having breast surgery.

DETAILED DESCRIPTION:
Study Groups:

If you are eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group.

If you are in Group 1, you will receive light electrical stimulation to the wrist area during surgery. You will also receive standard of care drugs to reduce PONV. If you have nausea or you are vomiting after surgery, you will receive additional standard of care drugs for those symptoms. You may ask the study staff for information about how the drugs are given and their risks.

If you are in Group 2, you will receive standard of care drugs to reduce PONV only (you will not receive electrical stimulation). If you have nausea or you are vomiting after surgery, you will receive additional standard of care drugs for those symptoms.

Electrical Stimulation:

The electrical stimulation is applied through a small sticky pad that is connected to a machine called a neuromuscular blockade monitor (NMBN). NMBNs are routinely used by anesthesiologists to monitor drug levels in muscles during surgery.

The pad will be placed on your wrist after you receive anesthesia and removed at the end of surgery so you will not know what group you are in.

Study Procedures:

Both Groups:

* You will have blood (about 2 teaspoons) collected intravenously (through your IV) during surgery. This blood will be used for genetic testing that may explain why people respond differently to treatments for nausea and vomiting.
* You will complete a questionnaire about your pre-treatment expectations and your nausea every 15 minutes after you wake up after surgery until you leave the clinic. It should take about 2-3 minutes to complete the questionnaire each time.

Length of Study:

Your participation in this study will be over once you leave the clinic after surgery.

This is an investigational study. The NMBM monitor is commercially available and FDA approved for use by anesthesiologists to monitor drug levels in the muscles during surgery. Its use in this study to control nausea/vomiting is investigational.

Up to 176 participants will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Adults at least 18 years of age
2. Female gender
3. History of patient reported PONV, CINV or motion sickness
4. Patients scheduled for Breast Surgery
5. Sign an informed consent indicating they are aware of the investigational nature of this study.

Exclusion Criteria:

1. Patients scheduled for paravertebral block
2. Upper extremity deformity contralateral to the site of disease that could interfere with accurate point location or alter the energy pathway as defined by traditional acupuncture theory
3. Local skin infections at or near the acustimulation site
4. Pre-existing nausea and vomiting, defined as nausea or vomiting requiring pharmacological treatment greater than 3 times in the week preceding screening
5. History of CVA or other central nervous system disorder resulting in residual weakness or paresis of extremity contralateral to the site of disease
6. Grade III or IV upper extremity peripheral neuropathy
7. Cardiac pacemakers. Patients involved in this protocol will receive electrical stimulation. For safety reasons, electrical stimulation should be avoided in patients with pacemakers
8. Metal implants for the treatment extremity. For safety reasons, use of electrical stimulation should be avoided
9. Current acknowledged use of any illicit drugs, medical marijuana (including Marinol), or evidence of alcohol abuse as defined by The American Psychiatric Association criteria. This includes patients who are currently in the recovery process.
10. Pregnancy as this would alter anesthesia plan
11. Bowel obstruction
12. Surgery that would not allow access to at least one P6 site.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia M. Kowalski, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period occurred between March 2016 to June 2018. 609 potential patients were identified from the breast surgery schedule and were approached to assess their interest in participation and eligibility screening, of which, 233 patients met eligibility criteria. Of these 233 eligible patients, 188 patients consented to the trial.
Pre-assignment Details: Of the 188 consented patients, 184 patients were randomized. Four consented patients were excluded from trial before randomization due to: One patient became ineligible after enrollment, one patient's surgery started before study preparation could be completed, and two patients found to be ineligible after enrollment.
Groups:
- Intervention: Anesthesiologist-provided intraoperative electrical stimulation of P6 with a neuromuscular blockade monitor, combined with prophylactic anti-emetics
- Control: Only prophylactic anti-emetics
Period: Overall Study
Arm/Group | Intervention | Control
Started | 92 | 92
Completed | 86 | 86
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Patient became ineligible after enrollment | 2 | 5
Not completed — Surgery started before study preparation could be completed | 0 | 1
Not completed — PACU data unable to be collected | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 86 | 86 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.41 (10.32) | 58.35 (11.71) | 57.88 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 86 | 172
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 13 | 29
  Not Hispanic or Latino | 69 | 71 | 140
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 9 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 71 | 64 | 135
  More than one race | 4 | 8 | 12
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 86 | 86 | 172

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Intervention to Prevent Post-Operative Nausea and Vomiting (PONV)
Description: Examine the efficacy of electrical stimulation of P6 combined with prophylactic anti-emetics versus pharmacological prophylaxis alone in preventing the incidence of PONV following breast surgery in patients at high-risk for PONV
  Complete control is defined as "No nausea≥3 & No vomiting & No use of anti-emetic during PACU stay"
Time Frame: During stay in post-operative anesthesia care unit, until discharge, an average of 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 86 | 86
Participants
  Fail | 19 | 12
  Success | 67 | 71
  Missing Information | 0 | 3
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.2787, Chi-squared

2. Secondary Outcome: Feasibility of Conducting Study
Description: Determine the study feasibility where feasibility is defined by at least 20% of screened patients meeting inclusion criteria ability, 50% of these patients consenting, and 75% of patients within the acupuncture study arm completing all procedures
Time Frame: At study consent and at PACU discharge
Population: Feasibility was defined in three different ways, and in accordance with each feasibility definition type, there was a different number of patients analyzed. Per protocol, for the "completed study" feasibility definition, we were only looking at the intervention arm. We were not looking at both arms.
Measure: Count of Participants; unit: Participants
Groups:
- Entire Study: Anesthesiologist-provided intraoperative electrical stimulation of P6 with a neuromuscular blockade monitor, combined with prophylactic anti-emetics (intervention) and participants only prophylactic anti-emetics (control)
Arm/Group | Entire Study
Number analyzed (Participants) | 609
Participants
  Screened eligible | 233
  Consented: number analyzed (Participants) | 233
  Consented | 188
  Completed study: number analyzed (Participants) | 92
  Completed study | 86

3. Secondary Outcome: Efficacy of Intervention to Prevent Need for Rescue Anti-emetics
Description: Examine the effects of intra-operative NMBM stimulation of P6 on whether or not any anti-emetics were used compared to the control group
Time Frame: During stay in post-operative anesthesia care unit, until discharge, an average of 1 day
Population: Number of participants analyzed does not match number of participants who completed in participant flow due to missing data
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 59 | 65
Participants
  No | 45 | 54
  Yes | 14 | 11
  0 | 45 | 54
  1 | 6 | 10
  2 | 7 | 1
  3 | 1 | 0

4. Secondary Outcome: Satisfaction
Description: Examine group differences in post-operative patient satisfaction with PONV management. Participants were asked to rate their satisfaction with their nausea and vomiting management on a scale of 0-10, where "0" equals "very dissatisfied", and "10" equals "extremely satisfied".
Time Frame: At discharge from post-operative anesthesia care unit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Satisfaction score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 83 | 76
Satisfaction score | 8.92 (2.51) | 9.25 (1.79)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.8252, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Efficacy of Intervention to Result in Decreased PACU Length-of-stay
Description: Explore if intra-operative NMBM stimulation of P6 results in decreased PACU length-of-stay
Time Frame: During stay in post-operative anesthesia care unit, until discharge, an average of 1 day
Measure: Mean (Standard Deviation); unit: number of minutes
Arm/Group | Intervention | Control
Number analyzed (Participants) | 86 | 83
number of minutes | 120 (53.07) | 119.46 (49.88)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.8277, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Expectancy
Description: Explore the associations between expectancy and response to P6 stimulation. Step 1 of 2 compares expectancy answers between groups. The expectancy questionnaire asks participants what their expectation is of the effects of the intervention on lowering their nausea after surgery, lowering their pain after surgery, enabling them to cope with nausea and/or pain better, and enabling them to have a better recovery after surgery. Possible answers are "Not at all agree", "A little agree", "Moderately agree", "Mostly agree", and "Completely agree".
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 86 | 86
Participants
  Response to ASES_Coping question: Not at all Agree/A little Agree | 13 | 8
  Response to ASES_Coping question: Moderately Agree | 14 | 18
  Response to ASES_Coping question: Mostly Agree/Completely Agree | 45 | 37
  Response to ASES_Coping question: Missing | 14 | 23
  Response to ASES_Nausea question: Not at all Agree/A little Agree | 11 | 6
  Response to ASES_Nausea question: Moderately Agree | 18 | 17
  Response to ASES_Nausea question: Mostly Agree/Completely Agree | 43 | 40
  Response to ASES_Nausea question: Missing | 14 | 23
  Response to ASES_Pain question: Not at all Agree/A little Agree | 17 | 17
  Response to ASES_Pain question: Moderately Agree | 18 | 18
  Response to ASES_Pain question: Mostly Agree/Completely Agree | 37 | 29
  Response to ASES_Pain question: Missing | 14 | 23
  Response to ASES_Recovery question: Not at all Agree/A little Agree | 14 | 10
  Response to ASES_Recovery question: Moderately Agree | 13 | 12
  Response to ASES_Recovery question: Mostly Agree/Completely Agree | 45 | 42
  Response to ASES_Recovery question: Missing | 14 | 23
Statistical Analysis 1: Comparison: Intervention vs Control; Response to ASES_Coping question (Re-categorized); Test type: Superiority; p = 0.3908, Chi-squared
Statistical Analysis 2: Comparison: Intervention vs Control; Response to ASES_Nausea question; Test type: Superiority; p = 0.6029, Chi-squared
Statistical Analysis 3: Comparison: Intervention vs Control; Response to ASES_Pain question; Test type: Superiority; p = 0.7785, Chi-squared
Statistical Analysis 4: Comparison: Intervention vs Control; Response to ASES_Recovery question (Re-categorized); Test type: Superiority; p = 0.8434, Chi-squared

7. Secondary Outcome: Expectancy and Response to P6 Stimulation
Description: Explore the associations between expectancy and response to P6 stimulation. Step 2 of 2 compares baseline expectancy answers and response to P6 stimulation outcome directly, without taking into account group assignment. The P6 stimulation outcome was categorized as "Fail" or "Success", where "Success" is defined as "No nausea≥3 & No vomiting & No use of anti-emetic during PACU stay".
Time Frame: During stay in post-operative anesthesia care unit, until discharge
Population: The statistical analysis was between expectancy response at baseline and response to P6 stimulation outcome of either fail or success during PACU stay until discharge, regardless of group assignment. Number of participants analyzed does not match number of participants who completed in participant flow due to missing data for the P6 stimulation outcome.
Measure: Count of Participants; unit: Participants
Groups:
- Fail: The P6 stimulation outcome was categorized as "Fail" or "Success", where "Fail" is defined as Nausea≥3 OR vomiting OR use of anti-emetic during PACU stay".
- Success: The P6 stimulation outcome was categorized as "Fail" or "Success", where "Success" is defined as "No nausea≥3 & No vomiting & No use of anti-emetic during PACU stay".
Arm/Group | Fail | Success
Number analyzed (Participants) | 31 | 138
Participants
  Response to ASES_Coping question: Not at all Agree/A little Agree | 6 | 15
  Response to ASES_Coping question: Moderately Agree | 6 | 25
  Response to ASES_Coping question: Mostly Agree/Completely Agree | 9 | 72
  Response to ASES_Coping question: Missing | 10 | 26
  Response to ASES_Nausea question: Not at all Agree/A little Agree | 5 | 12
  Response to ASES_Nausea question: Moderately Agree | 7 | 27
  Response to ASES_Nausea question: Mostly Agree/Completely Agree | 9 | 73
  Response to ASES_Nausea question: Missing | 10 | 26
  Response to ASES_Pain question: Not at all Agree/A little Agree | 7 | 27
  Response to ASES_Pain question: Moderately Agree | 5 | 30
  Response to ASES_Pain question: Mostly Agree/Completely Agree | 9 | 56
  Response to ASES_Pain question: Missing | 10 | 25
  Response to ASES_Recovery question: Not at all Agree/A little Agree | 7 | 17
  Response to ASES_Recovery question: Moderately Agree | 4 | 20
  Response to ASES_Recovery question: Mostly Agree/Completely Agree | 10 | 76
  Response to ASES_Recovery question: Missing | 10 | 25
Statistical Analysis 1: Comparison: Fail vs Success; Response to ASES_Coping question (Re-categorized) and P6 stimulation outcome; Test type: Other; p = 0.2742, Chi-squared
Statistical Analysis 2: Comparison: Fail vs Success; Response to ASES_Nausea question (Re-categorized) and P6 stimulation outcome; Test type: Other; p = 0.2747, Chi-squared
Statistical Analysis 3: Comparison: Fail vs Success; Response to ASES_Pain question (Re-categorized) and P6 stimulation outcome; Test type: Other; p = 0.5608, Chi-squared
Statistical Analysis 4: Comparison: Fail vs Success; Response to ASES_Recovery question (Re-categorized) and P6 stimulation outcome; Test type: Other; p = 0.1014, Chi-squared — There is no statistically significant association between expectancy and complete PONV control

ADVERSE EVENTS:
Time Frame: During stay in post-operative anesthesia care unit, until discharge, an average of 1 day
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/86
Other Adverse Events (participants affected / at risk) | 4/86 | 11/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=86) | Control (N=86)
Muscle weakness upper limb [left] (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle weakness upper limb [right] (Musculoskeletal and connective tissue disorders) | 0 | 3
Numbness in left arm (Nervous system disorders) | 1 | 2
Numbness in right arm (Nervous system disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Paresthesia [left] (Nervous system disorders) | 1 | 1
Paresthesia [right] (Nervous system disorders) | 0 | 1
Hematoma (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT02473042/Prot_SAP_001.pdf
  • Informed Consent Form (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT02473042/ICF_000.pdf